CLINICAL TRIAL: NCT02824848
Title: Comparison of Perception-Action Approach and Passive Stretching Interventions for Infants With Congenital Muscular Torticollis: A Single-Blind Randomized Clinical Trial
Brief Title: Perception-Action Approach vs. Passive Stretching for Infants With Congenital Muscular Torticollis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to COVID-19 pandemic and will not resume.
Sponsor: Rosalind Franklin University of Medicine and Science (Other)
Collaborators: Rady Children's Hospital, San Diego (Other)
Responsible Party: Principal Investigator, Mary Rahlin, Associate Professor, Rosalind Franklin University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 421 PT; 160161 (Other: UCSD Human Research Protections Program)
Record Dates: First submitted 2016-07-02; First posted 2016-07-07 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Congenital Muscular Torticollis
Keywords: congenital muscular torticollis; infants; passive stretching; perception-action approach
MeSH Terms: conditions — Congenital torticollis | interventions — Muscle Stretching Exercises; Range of Motion, Articular; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Passive Stretching (Active Comparator): Passive Stretching intervention components include static passive stretching, active assistive range of motion, assisted stretching of the involved cervical musculature, and associated strengthening activities aimed to elicit head righting in developmentally appropriate positions and during developmentally appropriate movement transitions. Intervention is progressed by increasing head tilt angles, duration of head righting, and frequency and number of repetitions.
  Interventions: Behavioral: Passive Stretching
- Perception-Action Approach (Active Comparator): P-A Approach intervention components include environmental set-up for activity and participation in play, and manual guidance in the form of light pressure applied to the infant's body in developmentally appropriate positions. Both components are designed to promote spontaneous exploration of the environment by the infant by suggesting small, incremental changes in his/her perceptual-motor orientation and contact with the support surface. Intervention is progressed by gradually removing environmental supports provided to the infant's body parts, and by removing the therapist's hands from the infant's body to allow for spontaneous exploration of a newly found contact with the support surface or new body configuration.
  Interventions: Behavioral: Perception-Action Approach

INTERVENTIONS:
Behavioral: Passive Stretching — Passive stretching and associated strengthening activities to change head/neck and body alignment
  Other Names: Passive movement, physical therapy
  Arms: Passive Stretching
Behavioral: Perception-Action Approach — Environmental set-up and gentle manual guidance to promote spontaneous exploration of alternative head/neck and body alignment possibilities
  Other Names: Perceptual-motor intervention, physical therapy
  Arms: Perception-Action Approach

SUMMARY:
Congenital muscular torticollis (CMT) results from tightness of neck musculature that causes the infant to tilt the head to one side and turn it to the other side. Infants with CMT also show unequal use of both sides of the body for movement and play. In this randomized clinical trial, researchers will compare two physical therapy (PT) treatment methods, passive stretching and Perception-Action (P-A) Approach, in their effects on head position and use of both sides of the body in infants with CMT. Behavior demonstrated during PT sessions by infants in the two groups will be also compared. Thirty-six infants with CMT will be randomly assigned to a passive stretching group or a P-A Approach group. The infants in both groups will attend 5 weekly PT sessions, including the initial evaluation, 3 subsequent weekly sessions, and a re-evaluation session. At visits 1 and 5, each infant's habitual head position, the ability to turn the head to both sides, muscle strength on both sides of the neck, motor development, and use of both sides of the body for movement and play will be assessed. Each infant's behavior exhibited during therapy will be assessed at visits 2-4. Results obtained from the two groups will be compared.

It is hypothesized that:

1. There will be significant gains achieved by both intervention groups between the initial and final assessments on the following outcome measures:

   1. Still photography
   2. Arthrodial goniometry used to assess active head rotation to both sides
   3. The Muscle Function Scale (MFS) used to assess neck muscle strength
   4. The Alberta Infant Motor Scale (AIMS) used to assess motor development
2. There will be no significant difference between the groups on the above listed measures after the intervention is completed.
3. The P-A Approach group will achieve greater gains than the passive stretching group between the initial and final assessments on the Functional Symmetry Observation Scale (FSOS) used to assess the use of both sides of the body for movement and play
4. The P-A Approach group will demonstrate higher Therapy Behavior Scale (TBS) scores than the passive stretching group assigned based on participants' behavior demonstrated during PT intervention sessions

DETAILED DESCRIPTION:
This prospective longitudinal study will be a two-group, single-blind, pre-post-test design randomized clinical trial (RCT). The purpose of this study will be two-fold:

1. To compare the efficacy of passive stretching and Perception-Action (P-A) Approach interventions in improving postural alignment, symmetrical use of both sides of the body during movement and play, and gross motor development in infants with congenital muscular torticollis (CMT)
2. To compare therapy-related behavior in infants with CMT undergoing passive stretching and P-A Approach interventions during physical therapy (PT) sessions

Within group comparisons will be made to assess change over time, and between group comparisons will be made to compare the effects of the two interventions. Both interventions are used in the clinic for infants with CMT but it is not known whether they are equally effective or if one is more effective than the other.

Thirty-six consecutively enrolled infants with CMT will be randomly assigned to a Passive Stretching group or a P-A Approach group using a blocked randomization procedure. Each infant will attend 5 weekly 60-minute PT sessions, including the initial evaluation, 3 interventions sessions, and a re-evaluation. The total duration of each participant's involvement in the study will be approximately 1-2 months. At visits 1 and 5, each infant's habitual head deviation from midline, active head rotation to both sides, neck muscle strength on both sides, motor development, and symmetrical use both sides of the body for movement and play will be assessed.

Participants' photos will be taken in a supine position and parts of the initial PT evaluation and re-evaluation sessions will be video recorded for future analyses by an assessor blind to the infants' group assignment. Such analyses will include still photography measurements, assessment of motor development using the Alberta Infant Motor Scale (AIMS), and assessment of symmetrical use of both sides of the body using the Functional Symmetry Observation Scale (FSOS). Treating therapists will perform "live" active head rotation and muscle strength measurements, for which assessor blinding will not be possible. In addition, each infant's behavior exhibited during therapy will be assessed by the treating therapist at intervention sessions 2-4. Results obtained from the two groups will be compared.

At the first PT visit, the treating therapist will conduct a PT evaluation, educate the caregiver in proper positioning and benefits of tummy time, and provide intervention specific to the infant's group assignment. For the Passive Stretching Group, intervention will include caregiver instruction in passive stretching for lateral flexion and rotation of the neck, with the parent practicing the techniques. For the P-A Approach Group, intervention will include the interpretation of the infant's behavior for the caregiver while manual guidance is provided to the infant. At 3 subsequent PT sessions, group-specific intervention and continued caregiver instruction will be provided. Passive Stretching Group intervention components will include passive stretching and associated strengthening activities. P-A Approach Group intervention components will include environmental set-up and manual guidance. At the final PT visit in the study, a PT re-evaluation will be conducted, followed by group-specific intervention as needed.

Prior to initiating the RCT, a pilot study will be conducted to establish the intrarater, test-retest or inter-rater reliability of the outcome measures, as appropriate. A total of 10 infants with CMT will be recruited for the pilot project.

Fidelity of intervention will be evaluated during the pilot study using a Fidelity of Intervention Checklist to ensure the treating therapists' adherence to the strategies outlined as essential elements of each of the intervention approaches. In addition, during the main study, intervention adherence will be assessed by tracking the participants' attendance, the PT session length and frequency, and the total duration of each subject's research participation.

ELIGIBILITY:
Inclusion Criteria:

* age between birth and 9 months at the time of recruitment
* diagnosis of congenital muscular torticollis as documented in the medical record
* Parents agree not to have their child participate in any additional interventions for CMT during the course of the study

Exclusion Criteria:

* other types of torticollis, such as neuromuscular torticollis, Sandifer syndrome, benign paroxysmal torticollis, ocular torticollis and other non-muscular types of torticollis, such as related to bony anomalies, which would warrant a referral back to the referring physician or to an appropriate specialist for diagnosis
* being seen for torticollis by another health care provider
* parents were using passive stretching with their infant prior to the study being offered to them AND would like to continue with passive stretching, but the child is assigned to the other intervention group
* parents were using Perception-Action Approach with their infant prior to the study being offered to them AND would like to continue with the same approach but the child is assigned to the other intervention group
* the child is found to meet the exclusion criteria at any time during the clinical trial

Max Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Still Photography | At baseline and week 5
  Change in the angle of habitual head deviation from midline assessed in a supine position
Arthrodial Goniometry | At baseline and week 5
  Change in the angular difference in active cervical rotation range of motion between the involved and uninvolved sides
Muscle Function Scale (MFS) | At baseline and week 5
  Change in the MFS score that reflects the difference in strength of lateral neck flexor muscles during head righting between the involved and uninvolved sides
Functional Symmetry Observation Scale (FSOS) | At baseline and week 5
  Change in the FSOS score that reflects functional use of both sides of the body during spontaneous movement and play
Alberta Infant Motor Scale (AIMS) | At baseline and week 5
  Change in the AIMS score that reflects gross motor development while also considering symmetrical postural alignment and symmetrical use of both sides of the body during movement and play

SECONDARY OUTCOMES:
Therapy Behavior Scale (TBS) | Weeks 2, 3 and 4 (at the time of intervention sessions 2, 3 and 4)
  The TBS score documents therapy-related behavior during intervention sessions; to be used for between group comparison only.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Rahlin, PT, DHS, PCS, Principal Investigator — Rosalind Franklin University of Medicine and Science; Nancy Haney, PT, MS, Principal Investigator — Rady Children' Hospital, San Diego
Locations (1):
- Rady Children's Hospital, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Kaplan SL, Coulter C, Fetters L. Physical therapy management of congenital muscular torticollis: an evidence-based clinical practice guideline: from the Section on Pediatrics of the American Physical Therapy Association. Pediatr Phys Ther. 2013 Winter;25(4):348-94. doi: 10.1097/PEP.0b013e3182a778d2. PMID 24076627
- [Background] Rahlin M. TAMO therapy as a major component of physical therapy intervention for an infant with congenital muscular torticollis: a case report. Pediatr Phys Ther. 2005 Fall;17(3):209-18. doi: 10.1097/01.pep.0000179176.20035.f0. PMID 16357675
- [Background] Cheng JC, Chen TM, Tang SP, Shum SL, Wong MW, Metreweli C. Snapping during manual stretching in congenital muscular torticollis. Clin Orthop Relat Res. 2001 Mar;(384):237-44. doi: 10.1097/00003086-200103000-00028. PMID 11249171
- [Background] Tscharnuter I. Clinical Application of Dynamic Theory Concepts According to Tscharnuter Akademie for Movement Organization (TAMO) Therapy. Pediatr Phys Ther. 2002 Spring;14(1):29-37. PMID 17053679
- [Background] Ohman A, Nilsson S, Beckung E. Stretching treatment for infants with congenital muscular torticollis: physiotherapist or parents? A randomized pilot study. PM R. 2010 Dec;2(12):1073-9. doi: 10.1016/j.pmrj.2010.08.008. PMID 21145518
- [Background] Rahlin M, Sarmiento B. Reliability of still photography measuring habitual head deviation from midline in infants with congenital muscular torticollis. Pediatr Phys Ther. 2010 Winter;22(4):399-406. doi: 10.1097/PEP.0b013e3181f9d72d. PMID 21068640
- [Background] Blanchard Y, Neilan E, Busanich J, Garavuso L, Klimas D. Interrater reliability of early intervention providers scoring the alberta infant motor scale. Pediatr Phys Ther. 2004 Spring;16(1):13-8. doi: 10.1097/01.PEP.0000113272.34023.56. PMID 17057466
- [Background] Rahlin M, McCloy C, Henderson R, Long T, Rheault W. Development and content validity of the Therapy Behavior Scale. Infant Behav Dev. 2012 Jun;35(3):452-65. doi: 10.1016/j.infbeh.2012.03.001. Epub 2012 Jun 26. PMID 22729134